<u>Official Study Title:</u> A Phase I, First-in-Human, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study of the Safety and Efficacy of Allogeneic Mesenchymal Stem Cells in Cancer Survivors with Anthracycline-Induced Cardiomyopathy

**Short Title**: Stem Cell Injection in Cancer Survivors (SENECA)

NCT: NCT02509156

**<u>Date of Informed Consent Document</u>**: IRB approval date 06/13/2017

Protocol Title: A Phase I, First-in-Human, Multicenter, Randomized, Double-Blinded,

Placebo-Controlled Study of the Safety and Efficacy of Allogeneic Mesenchymal Stem Cells in Cancer Survivors with Anthracycline-

**Induced Cardiomyopathy** 

(<INSERT IRB APPROVAL NUMBER HERE>)

Study Identifier: SENECA

Study Sponsor: The Cardiovascular Cell Therapy Research Network (CCTRN)

Principal Investigator: <Insert INVESTIGATOR NAME HERE>

<INSERT INVESTIGATOR INSTITUTION HERE>

#### INVITATION TO TAKE PART

You are being invited to take part in a research study (title above) conducted by <INVESTIGATOR NAME> and his/her staff at <INSTITUTION NAME>. This is a national study with six other centers located across the country. The study will enroll approximately 36 people nationally. This location will enroll approximately 8-10 people.

This study has funding from The National Heart, Lung, and Blood Institute (NHLBI), which is part of the National Institutes of Health. This research study has been reviewed by the <INSERT NAME OF IRB and IRB APPROVAL NUMBER>.

Your decision to take part is voluntary and you may refuse to take part, or choose to stop taking part, at any time during the study. A decision not to take part or to stop being a part of this research study will not change the healthcare services that are available to you by the doctor, hospital, or other clinics.

You may refuse to answer any questions asked or written on any forms.

The nature of the study, benefits, risks, discomforts, and other information about the study are discussed below. You will be told of any findings discovered during the study, which may affect your willingness to take part. You are urged to discuss any questions you have, about the study, with the research staff.

<INSERT INVESTIGATOR CONFLICT OF INTEREST INFORMATION HERE IF APPLICABLE>
One or more of the investigators conducting this study serve as paid speakers, consultants or advisory committee members for a company that makes or promotes products used in this study. These financial interests are within permissible limits established by the <Institution Name> Conflict of Interest Policy. If you have any questions regarding conflicts of interest, please ask your study doctor or call the Institutional Review Board at <INSERT PHONE>

### PURPOSE AND BACKGROUND INFORMATION

Common use of a group of cancer medications called anthracyclines has dramatically improved cancer survival numbers over the past 50 years. Anthracycline-based cancer medications remain common and effective treatments for breast cancer, lymphomas, leukemias, and sarcomas. Unfortunately, the use of anthracyclines is limited due to their poisonous effects on the heart, including the development of a form of heart failure called anthracycline-induced cardiomyopathy (AIC). These effects can be seen as late as

gRB NUMBER: HSC-SPH-15-0443 UTHealth IRB APPROVAL DATE: 06/13/2017 20 years after the cancer treatment. Current treatments for AIC reduce the symptoms but there is no cure for this disease. While studies suggest that the usual medications used to treat heart failure (e.g. ACE inhibitors, angiotensin receptor blockers, beta-blockers, and statins) may help treat AIC, there continues to be a group of patients that will develop worsening symptoms and end-stage heart failure despite the best medical therapy, with many individuals worsening to the point of requiring a heart transplant. Due to the small number of donor organs, very few people receive heart transplants when they need one.

Stem cells are cells that do not yet have a specific function in the body. Mesenchymal stem cells (MSCs) are a type of stem cell that can be grown from bone marrow (the spongy tissue inside of bones). Stem cells can develop into other types of more mature (specific) cells, such as blood and muscle cells. It is hoped that by placing these cells into your heart, they will allow the heart to work better and reduce the scarred heart tissue associated with heart failure.

Rather than taking these cells from your own bone marrow (which has been exposed to the cancer medications in the past), MSCs can be taken from a healthy donor (who has never had chemotherapy). This type of stem cell is called allogeneic (or allo for short).

The purpose of this research study is to determine whether giving allo-MSCs to patients with AIC is safe and whether these treatments improve heart function. You are being asked to be in this research study because you have been diagnosed with AIC and you have been cancer-free for at least two years. You also have left ventricular dysfunction (your heart does not pump blood as well as it should) and because of this you are experiencing heart failure.

### Randomization

If you agree to take part in this study, you will be randomized (similar to flipping a coin) to receive one of two study products: allo-MSCs or a placebo (which is a solution that contains no cells, only salt and proteins). It is not known whether the cells will be of benefit. For this reason, some study participants must receive a placebo. This will allow a careful comparison to study the benefits and side effects of the study product containing cells. One half of the patients will receive allo-MSCs and one half of the patients will receive placebo. Neither you nor your doctors treating you will know what study product you will receive. Regardless of which group you are in, you will otherwise receive the same standard treatment for your heart failure.

The allo-MSCs given to you in this study will be taken from the bone marrow of a healthy human donor. Giving patients allo-MSCs, is an investigational procedure that has been authorized by the Food and Drug Administration (FDA) for this study.

### STUDY PROCEDURES AND ASSOCIATED RISKS

Importantly, your taking part in this research study will not affect the usual treatment of medical therapy that all patients with heart failure receive. If you agree to take part in this study you will undergo several tests and procedures during outpatient visits and during the follow-up visits which are in addition to those normally performed for patients being treated for heart failure. To take part in this study, you must return for all scheduled follow-up visits, as instructed by your doctor, until follow-up is no longer necessary. As a participant in this study, you agree to keep your doctor informed of all future changes in your address and phone number.

After you sign the informed consent form, you will be asked to have several tests and exams to see if you are eligible for the study. You will have up to 45 days to complete these tests, depending on the schedule you work out with your study doctor. It is possible that after you have completed these tests, the results

UTHealth IRB APPROVAL DATE: 06/13/2017

may show that you do not qualify for the study. This means you would not be eligible to receive the study product. If this happens, you will be informed of the reason(s) you are not eligible and will be referred back to your regular doctor for care.

A schedule and brief descriptions of the research activities are provided below.

## **Schedule of Study Visits**

# **Baseline Visit (approximately 6 hours)**

| TEST | TIME for TEST (approximate) |
|---|---|
| Discuss and Sign Consent Form | 45 minutes to 1hour |
| History and Physical Exam | 45 minutes |
| Questionnaire | 20 minutes |
| ECG | 30 minutes |
| Labs-Blood work | 15 minutes |
| Pregnancy test (females) | 10 minutes |
| Exercise Testing (six minute walk)- two tests* | 45 minutes each |
| MRI (with ICD evaluation) | 1-1.5 hours |
| Stress echocardiogram (NOT ALL PARTICIPANTS)** | 30 minutes |

<sup>\*</sup>A third test may be required depending on results from the first two tests.

# **Study Product Injection Visit (approximately 3-3.5 hrs)**

| TEST | TIME for TEST (approximate) |
|----------------------------------------|-----------------------------|
| Physical Exam | 30 minutes |
| ECG | 30 minutes |
| Labs-Blood work | 15 minutes |
| Pregnancy test (females) | 10 minutes |
| Blood draw-biorepository only | 15 minutes |
| ICD evaluation (if applicable) | 10 minutes |
| Cardiac Catheterization/NOGA procedure | 1 hour |
| Echocardiogram | 30 minutes |

# Day after Injection Visit (approximately 1.5 hrs)

| TEST | TIME for TEST (approximate) |
|-------------------------------|-----------------------------|
| Physical Exam* | 30 minutes |
| ECG | 30 minutes |
| Labs- Blood work | 15 minutes |
| Blood draw-biorepository only | 15 minutes |

<sup>\*</sup>Patient receives temperature log to monitor for infection.

## One week Follow Up (approximately 1.5 hrs)

| TEST | TIME for TEST (approximate) |
|-------------------------------|-----------------------------|
| Physical Exam | 30 minutes |
| ECG | 30 minutes |
| Labs-Blood work | 15 minutes |
| Blood draw-biorepository only | 15 minutes |

<sup>\*\*</sup> Only participants who have no available imaging in the last 5 years

## One month Follow Up (approximately 1 hr)

| TEST | TIME for TEST (approximate) |
|-------------------------------|-----------------------------|
| Physical Exam | 30 minutes |
| Labs-Blood work | 15 minutes |
| Blood draw-biorepository only | 15 minutes |

# Six month Follow Up (approximately 4.5-5 hrs)

| TEST | TIME for TEST (approximate) |
|---|---|
| Physical Exam | 30 minutes |
| Questionnaire | 20 minutes |
| ECG | 30 minutes |
| Labs- Blood work | 15 minutes |
| Pregnancy test (females) | 10 minutes |
| Blood draw-biorepository only | 15 minutes |
| MRI (with ICD evaluation) | 1-1.5 hours |
| Exercise Testing (six minute walk)- two tests* | 45 minutes each |

<sup>\*</sup>A third test may be required depending on results from the first two tests.

## Twelve month Follow Up (approximately 4.5-5 hrs)

| TEST | TIME for TEST (approximate) |
|---|---|
| Physical Exam | 30 minutes |
| Questionnaire | 20 minutes |
| ECG | 30 minutes |
| Labs- Blood work | 15 minutes |
| Pregnancy test (females) | 10 minutes |
| MRI (with ICD evaluation) | 1-1.5 hours |
| Exercise Testing (six minute walk)- two tests* | 45 minutes each |

<sup>\*</sup>A third test may be required depending on results from the first two tests.

# **Telephone Contact- Twenty-four month Follow Up (approximately 20 minutes)**

| ACTIVITY | TIME for ACTIVITY (approximate) |
|---------------------|---------------------------------|
| Telephone Interview | 20 minutes |

# Descriptions of Research Activities

### **History and Physical Exam**

Your medical history and current use of medicines will be reviewed. You will also undergo a physical exam which will include temperature, blood pressure, heart rate, and breathing rate, as well as height and weight measurement.

#### **ECG**

An electrocardiogram (ECG) is a tracing of your heart rhythm and is used to record the electrical activity of your heart. These will take place during six of your visits.

#### Labs

A needle will be inserted into the vein of your arm and blood will be withdrawn (about 2-3 tablespoons on seven different occasions or about 14-21 tablespoons total for the entire trial). If you agree to the optional biorepository (described later in this consent form) there will be additional blood draws on five occasions.

As required by the cell processing facility and the Food and Drug Administration (FDA), your blood will be tested for certain viruses such as hepatitis and HIV. If you test positive for active Hepatitis B, Hepatitis C, or HIV you will not be able to take part in this study. In addition, the lab is required by law to report positive results to <INSERT ALL RELEVANT STATE REPORTING AGENCIES>. Reportable data may include: patient name, birth date, ethnicity, race, residence, date of specimen collection, treatment prescribed or dispensed, treatment date, doctor name, address, phone number, and other information related to the case. You will also be told of a positive HIV or Hepatitis B or C test.

## The Minnesota Living with Heart Failure Questionnaire

This questionnaire asks how your daily activities (such as job, family life, and food habits) are affected by your condition. This questionnaire will take about 15 minutes to fill out. You will also be asked these questions during the baseline period and follow-up appointments at months 6 and 12.

### Six Minute Walk Test

You will be asked to walk in a corridor (without elevation). You will be asked to walk at your own pace, while trying to cover as much ground as possible in six minutes. You can stop and rest during the test, but you will be asked to resume walking as soon as you feel you are able to do so. After six minutes, you will be asked to stop walking. The total distance walked and symptoms experienced during the walk (e.g., chest pain, trouble breathing, a feeling of tiredness, dizziness) will be recorded. This testing will be completed at the beginning of the study and also at months 6 and 12. At each of these visits you will complete this test twice, with time in between the tests for you to rest. In rare circumstances, you may be asked to complete the test a third time, depending on the results of the first two tests

#### MRI and ICD Evaluation

You will have a **Magnetic Resonance Imaging (MRI)** exam at the beginning of the study and again at the 6- and 12-month visits. A MRI is used to determine how healthy your heart is and how well it works. MRI uses large magnets and radio frequency waves to make pictures of the inside of the body; no radiation exposure is involved. This test gathers information about the heart by creating moving images of the heart while it is beating. The MRI is used to look at the presence of disease in the heart.

Before this test, you will be asked if you have certain metals in your body. Additionally, **if you have a pacemaker/internal cardiac defibrillator (ICD)**, the study doctor will check your device by using a wand placed on the skin over your ICD. The study team will be checking you during the test by using a blood pressure cuff, heart monitor, and oxygen monitor throughout the scan. The MRI scans take 60-90 minutes on average, but may take a little longer (20-30 additional minutes) if you have one of these devices.

During your MRI exam, you will lie on a padded table. You will have an intravenous (IV) line placed in your arm. A soft padded coil will be placed at the area where the pictures will be taken. The coil is necessary to help the MRI machine take pictures. The table will be moved into the center of a long narrow tube. If you have a history of claustrophobia (being uncomfortable in an enclosed space), tell the study nurse in advance. A small dose of medicine <INSERT NAME OF MED HERE> can be given to help you feel less anxious. A large magnet inside the tube will begin taking pictures. When the pictures are taken, it is normal for the MRI machine to make loud banging and clicking noises. You may be asked to wear earplugs or headphones for your comfort during the exam. During the exam, the MRI staff is able to see and hear you and you can hear the MRI staff. The MRI staff will be talking to you throughout your

UTHealth IRB APPROVAL DATE: 06/13/2017

MRI exam and may give you simple instructions, such as to hold your breath. You will be asked to lie perfectly still throughout the exam. At some point during the exam the MRI staff will stop the scanning procedure in order to put a contrast dye into a vein in the IV line in your arm. The contrast dye makes the heart more visible in the pictures.

## Cardiac Catheterization/Left Ventricular Angiocardiography and NOGA Mapping

During this procedure for the study, the doctor will insert a long, narrow tube called a catheter, into a blood vessel, usually in your leg, and then guide the catheter to your heart with the help of a special X-ray machine. X-ray dye is then injected through the catheter so that the X-ray machine can take pictures/movies of the left ventricle (left lower chamber) of your heart. The doctor uses a special device, called NOGA, which monitors the electrical and mechanical function of your heart. This procedure, referred to as NOGA mapping, will help your doctor find out which part of your heart muscle is still healthy but is not receiving enough blood and oxygen because this is the part that is most likely to respond to the study product injections. This helps the doctor decide where to inject the study product.

# **Study Product Injection**

Your doctor will use a special catheter with a retractable needle (called a NOGA Myostar catheter) to inject the study product into the damaged area of your heart muscle. This catheter is investigational and not approved by the FDA. There will be about 20 injections of a very small amount (a drop) of fluid containing millions of cells, or placebo, into your heart muscle. Following the procedure, you will be watched carefully, overnight in a telemetry (ECG monitored) unit.

## **Echocardiogram (Echo)**

An echocardiogram (echo) is an ultrasound image of your heart. It is used to see how well your heart is working. First a gel is put on your chest. A device called a transducer is moved over the surface of your chest. The transducer picks up the sound waves from your heart and sends them to a monitor to show a picture. This test checks the heart size, how well it pumps, and how well the heart valves look and work. There is no exposure to radiation with this test. A dye that helps the echocardiogram device to look at your heart may be injected into one of your veins as part of this procedure. You will have an echo after the study product injection, during the hospitalization period of the study.

## Stress Echocardiogram (Stress echo)- (NOT ALL PARTICIPANTS)

During this test, an echocardiogram is done both before and after your heart is stressed either by having you exercise or by injecting a medicine that makes your heart beat harder and faster (to imitate exercise). A stress echocardiogram is usually done to find out if you might have decreased blood flow to your heart (coronary artery disease). You would only have this test done if the study physician thinks you may have coronary artery disease and there are no recent tests in your medical record that test for it.

### **Temperature Log**

You will be asked to take and record your temperature two times a day for one week following your injection procedure. The purpose of this is to monitor for infection. You will be given a "Temperature Log" before you are discharged to keep track of your temperatures twice a day for 1 week. Instructions for reporting an increase in temperature are on the log. You will be asked to turn in your log at your one-week visit. Should signs of infection be present, your study doctor will ask you to return for a physical examination, and if necessary you may be started on an antibiotic treatment.

### **FOLLOW-UP EVALUATIONS**

### **Follow up Visits**

You will be asked to return for follow-up visits at 1 week and 1-, 6- and 12 months after your injection procedure. A brief telephone interview will be conducted at 24 months. Please refer to the schedule of activities for specifics tests and assessments to be performed at each visit.

#### **Time Commitment**

The study elements and time are: (1) <u>Baseline testing and injection visits</u>- about 9 hours over several days; (2) <u>overnight stay following injection and day of discharge activities</u> (about 24 hours); (3) <u>follow up visit procedures</u>- includes four follow up appointments at 1 week and 1, 6, and 12 months after the injection procedure (range from 1-5 hours each, 12-15 hours total); and (4) <u>follow up telephone interview at 24 months</u> (about 20-30 minutes). **The total maximum number of hours is about 49 hours**.

### **ALTERNATIVES**

You may choose not to participate in this study. Alternative forms of therapy exist for patients who have chronic heart problems. If you choose not to take part, you can receive the standard therapy for people who are experiencing heart failure symptoms. Optimal medication management would be the most common alternative therapy for you.

### RISKS AND/OR DISCOMFORTS

Your doctor will explain all the possible risks of the procedures associated with this study. The specific risks and discomforts for each test are described below. As with any procedure, whether it is investigational or approved, there may be risks which are unanticipated or unknown at this time.

#### **ECG**

It may be necessary to shave small areas of your chest to apply the adhesive patches. You may experience slight discomfort when the adhesive patches are removed.

#### Labs

Risks associated with drawing blood from your arm include pain, bruising, site swelling, light-headedness and, on rare occasions, infection.

**Special note to women:** Being part of this study while pregnant may expose the unborn child to significant risks, some of which may be currently unforeseeable. Therefore, pregnant women will be excluded from the study. If you are a woman able to become pregnant, a pregnancy test will be done and it must be negative before you can continue in this study. If sexually active, you must agree to use appropriate contraceptive measures while taking part in this study. Medically acceptable contraceptives include: (1) surgical sterilization (such as tubal ligation or hysterectomy), 2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) intrauterine device (IUD). If you become pregnant while taking part in this study or if you have unprotected sex, you must inform the study doctor immediately.

### **Questionnaire**

Some of the questions on the questionnaire ask you to consider areas of your life which you may not commonly think about. There are no physical risks from completing the survey, but the questions could cause you concern or possibly emotional distress.

## **Exercise Testing (Six minute walk test)**

During this test, you may experience episodes of temporary lightheadedness, fainting, chest discomfort, leg cramps, and very rarely, heart attack.

## Stress Echocardiogram (NOT ALL PARTICIPANTS)

Only participants who have no other available imaging in their recent medical history will have this test. This test simulates the how the heart works during exercise. Due to that, you may feel a sense of extreme tiredness, temporary irregular heartbeat, dizziness, nausea, high blood pressure, chest pain, and in very rare circumstances heart attack.

## Magnetic Resonance Imaging (MRI) procedure

There may be mild to moderate risks and discomforts with placement of an IV line, administration of medications, or the blood draw. The risks of starting an IV and drawing blood include pain, redness, minor bleeding, swelling, and bruising at the injection site. Rarely, lightheadedness, fainting, and infection might happen. The nurse will monitor you and appropriate treatments will be given if you develop any complications.

You may feel uncomfortable or tired from lying down in the MRI machine. You will be asked to hold your breath. Each breath hold lasts about 10-15 seconds. If you are anxious or have a history of claustrophobia (feeling uncomfortable in small enclosed spaces), you may experience this during the MRI; as noted above, medication can be made available to help you relax. Administration of contrast dye may cause nausea, vomiting, or headache. Allergic reactions to contrast dye are rare, but there are extremely rare instances of reactions causing death.

The contrast dye used in the cMRI procedure is referred to as a gadolinium based contrast agent (GBCAs). After it is given, GBCAs leave the body mostly through the kidneys. Recent medical papers report some deposits from GBCAs remain in the brains of some patients who have four or more contrast MRI scans, long after the last dose is received. Recent studies conducted in humans and animals have confirmed that these deposits can remain in the brain, even in people with normal kidney function. It is unknown whether these deposits are harmful or can lead to adverse health effects. Available information does not identify any adverse health effects. However, this issue continues to be studied by the FDA and you will be informed should any new specific danger or threat to your health emerge.

The contrast dye may also induce kidney damage or nephrogenic systemic fibrosis (NSF), a serious and potentially fatal disease that involves the skin, muscle, and internal organs. The risk of this is increased with patients who already had some evidence of kidney disease or diabetes, or are dehydrated. In general, if a patient has normal kidney function, then the risks of kidney failure caused by contrast dye are small. Your kidneys will be tested prior to any dye that would be given. You should contact your doctor if you develop signs or symptoms of NSF, which include: Skin burning or itching, reddened or darkened patches and/or skin swelling, hardening and/or tightening; yellow raised spots on the whites of the eyes; joint stiffness, limited range of motion in the arms, hands, legs or feet; pain deep in the hip bone or ribs; and/or muscle weakness.

There is no radiation (x-ray) exposure from MRIs. There is a risk of heat injury from radiofrequency coils and the cables to the coil and monitoring equipment (heart monitor, oxygen monitor, etc.). Please report any heating or burning sensation immediately and the scan will be stopped.

For those with pacemakers and ICDs: Magnetic resonance imaging works by generating a strong magnetic field. Both pacemakers and ICDs are devices that contain wires with electrodes that are connected to one or more of your heart's chambers. These are designed to restore normal rhythm to the heart by sending electrical pulses through the wires. It is important that you know that some, but not all, of these devices are approved by the FDA to be used in a MRI scanning environment. Researchers have imaged hundreds of patients with such devices under careful monitoring without incident. The investigators of this study have undergone training in these imaging techniques and will follow the best safety practices from these researchers. The powerful magnetic fields and radio waves that are part of MRI scans could cause the ICD wires to overheat, potentially damaging heart tissue. MRIs can induce unwanted currents that would either make the heart beat wildly, or in the case of ICDs, cause an unnecessary shock.

Pacemakers and ICDs can be temporarily reprogrammed so they don't react to an MRI's magnetic field. Reprogramming a pacemaker or ICD can be done noninvasively through the skin with a wand like device. Pacemakers can be put into the "inhibited pacing mode," which means the heartbeat has to get very slow before the device activates and starts helping the heart beat regularly. The part of the ICD that senses a racing, irregular heartbeat (tachycardia) is temporarily disabled.

If you have a pacemaker/ICD, it will be monitored during the MRI scan. Theoretically, the MRI scan could interfere with, or possibly damage, your pacemaker/ICD, but its functioning will be verified immediately after the procedure. During the scan you are at an increased risk of experiencing an arrhythmia, which could be life threatening or fatal (result in death). A cardiologist or trained registered nurse with pacemaker/ICD expertise will check your device before, during, and after the scan to ensure your safety. Trained life support staff will be present and a crash cart (defibrillator) will be available during the procedure should you experience a life threatening arrhythmia. The staff will keep in contact with you visually and vocally throughout the procedure. You will be monitored continuously during the scan.

### **Cell Processing Procedure**

If you happen to receive the allo-MSC cell product, it is possible that your body might react and reject the allo-MSC cells. Human clinical research studies with allo-MSCs in heart patients have provided evidence against the occurrence of rejection of the transplanted cells and also against the occurrence of graft versus host disease (GVHD), where healthy infused cells recognize the tissues of the person receiving the cells as "foreign" and mount an immunologic attack.

Processing the cells is done under strict sterile conditions; however, there is a rare chance that the cells could get contaminated while being processed. Testing will be done on the cells; however, it takes about 2 weeks to get the final results. If the tests show your cells were contaminated, you will be notified and instructed on whether or not you should be treated with antibiotics. You will be taking your temperature twice a day for one week, which may help determine if you are developing an infection before the test results are known.

There may be some circumstances where we are unable to give you the processed cells; such as a processing failure or poor quality of the cells. If events such as these occur, you will not receive the allo-MSC cells but we will ask you to continue with follow up in the study as already discussed. Processes in place to prevent these failures include: the use of standard operating procedures for preparing the allo-MSC cell product, which will identify any problems with the study product before it is released, and continuous temperature monitoring of the product during shipment to the hospital at which you will receive them.

## **Mapping and Injection Procedures**

### **Anticoagulation Medications**

If you are taking anticoagulation medications (i.e. blood thinners) at the time of the mapping and injection procedures, some of these medications (e.g. Coumadin) may be stopped for a short period before the procedures; during which time you may be at an increased risk of a stroke. It is very important that you inform the research team immediately of any symptoms of dizziness, light-headedness, blurred vision, slurred speech, facial drooping, decrease sensations anywhere on your body, or weakness or a decrease in strength of your arms or legs. You will be closely monitored, during any interruption in anticoagulation therapy, for the events listed above.

# Cardiac Catheterization and NOGA Mapping

Your study doctor will fully explain this procedure and associated risks to you. Some problems that might happen include (but others could occur) oozing of blood around where the catheter (small hollow tube) goes into your skin, a swelling filled with blood (hematoma) under the skin, allergic reaction to the dye that is injected when the doctor looks at the heart vessels (angiography) either during or following the study product injection procedure, or formation of a blood clot (a blockage) at the place where the catheter goes into your skin. A blood clot could stop the flow of blood or hurt the blood vessel. If blood flow is stopped or slowed a lot, the body parts that rely on that blood could also be damaged, which could lead to loss of function or surgical removal of the body part, or could worsen your heart condition and its symptoms. Other problems that could happen because of this test are: local nerve damage (loss of feeling), infection, changes in the how your heart beats, stroke, and heart attack. Some temporary problems that might happen are: temporary movements (spasm) of a muscle, vein, or artery; pulling apart of blood vessel walls (separation of the layers of the walls of a blood vessel); or sudden blockage (closure) of a blood vessel. A very rare complication could result in death or a need for an urgent coronary artery bypass graft (open heart surgery). Serious complications, including death, happen in less than 1 in every 1,000 tests that are performed.

The risks of the use of the iodine that is in the contrast media for the heart angiography procedure are rare. Some problems that might occur are hypersensitivity or even severe allergic reactions, or decreased kidney function, particularly if you have underlying kidney problems. Your doctor will measure your kidney function before this procedure to find out if your kidneys are working properly.

The possible risks of NOGA mapping include, but are not limited to: damage to blood vessels, bleeding, infection, inflammation of the sac surrounding the heart, damage to kidneys, a small risk of heart attack, stroke, damage to the heart valves, perforation (a small hole) in the heart causing blood to accumulate around the heart, irregular heartbeats (including ventricular tachycardia and ventricular fibrillation), possible ICD firing, decreased blood pressure, dislodgement of material into other arteries leading to possible blockage, radiation exposure and a very small risk of death. You will receive some radiation as part of the NOGA study (see the Radiation Risks Section below).

# **Study Product Injection**

The catheter used to inject the study product is investigational (not yet approved for this use by the FDA). Some problems that might happen include (but others could occur): decreased blood pressure, irregular heartbeats, possible firing of ICD, chest pain or discomfort, damage to the heart muscle, perforation of the heart causing blood to accumulate around the heart, bleeding, heart attack, stroke, dislodgement of material into other arteries (possibly causing blockage), need for emergency surgery such as coronary re-vascularization, and death. It is possible that a small amount of cells will enter the bloodstream of the heart rather than the heart muscle. If the injection catheter penetrates through the heart (from inside to outside) and cells appear in the fluid filled area surrounding your heart, which

IRB NUMBER: HSC-SPH-15-0443 UTHealth IRB APPROVAL DATE: 06/13/2017 cushions the heart as it moves (pericardial space) there is a possibility of potentially harmful effects which could cause an inflammatory response. Injection directly into the heart muscle also may cause inflammation or irritability. Your medical team will closely monitor you to minimize the chance of any problems occurring during the procedure.

# **Radiation Risks**

The mapping/injection procedure involves exposure to radiation, which is in addition to what you may receive as part of your standard care. The benefit from the radiation you receive for your standard care typically outweighs the risk because it allows your doctor to provide appropriate medical care; however, the additional radiation "dose" you receive for research purposes may not benefit you personally. There are established annual radiation dose limits for both individuals who work with radiation (e.g. x-ray technologists, radiologists, etc.) and those participating in research studies. The additional radiation dose you will receive from participating in this study is less than either of those limits.

Radiation has been shown to cause cancer and/or leukemia from doses that are significantly higher than the additional annual radiation dose you will receive by participating in this study. According to the Health Physics Society (an international organization that specializes in radiation protection), the increased risk of health effects (i.e. cancer and/or leukemia) from radiation doses of this amount is either too small to be observed or nonexistent in a normal population. While there is no evidence that any risk exists for humans exposed to such low levels, it is assumed that the risks rise with lifetime accumulated dose from all sources of ionizing radiation, including the doses you receive from medical procedures and the environment. You should also be aware that everyone's sensitivity to radiation is not the same and some diseases (e.g. genetic diseases, diseases affecting DNA repair, and immune diseases such as HIV) may make you more sensitive to the effects and consequences of the radiation exposure than the normal population. Finally, you should know that even if there is an increased risk of an effect, it could be 5 to 20 years before any effect would actually occur. Thus, you may want to factor in your age, overall health, and the number of medical radiation procedures that you've had when determining if this risk is acceptable to you. The calculated effective dose resulting from your participation in this study is available upon request.

### **Risks That Are Not Known**

Because cell therapy treatment is investigational, that is not FDA approved, there may be risks that we do not know about at this time. There are no long-term safety data available. If we discover new risk information during the study, we will share this information with you.

Participation in more than one research study or project may further increase the risk to you. If you are already enrolled in a research study, please tell the person reviewing this consent with you before enrolling in this or any other research study or project.

### **BENEFITS**

It is not known whether this procedure is beneficial. It may improve the way your heart muscle functions. This may also help with daily activities (e.g. walking for longer periods without symptoms) which may improve the quality of your daily life. The information gained from the research study will help answer these questions, not only for you but, for the general population. It is also possible that you may not receive any direct benefit from this research study. The information learned in this research study may help researchers better understand how safe it is to use stem cells in the heart and may help advance medical knowledge in general.

### WITHDRAWAL

You may withdraw your consent to take part in this study at any time. If you choose to withdraw from the study you will receive the usual standard of care without any loss of healthcare services. Also, your doctor may end your participation if continuing in the study does not appear to be in your best medical interest. <INSERT INVESTIGATOR NAME HERE>may end your participation in the study at any time. If you decide to withdraw from the study, your data collected prior to withdrawal may still be used up to the point of withdrawal.

Your doctor or the sponsor can stop the study at any time for any of the following reasons: if you have an adverse effect from the study drugs, if you need a treatment not allowed in this study, if you are unable to keep your appointments with your doctor, if you do not take the study drug as instructed, if you do not later consent to future changes that are made in the study plan, if the study is stopped by the FDA or the sponsor ahead of schedule, or for any other reason. Should the study be stopped, your study doctor will discuss other options with you.

### **CONFIDENTIALITY**

Please understand that representatives of the Food and Drug Administration (FDA), the <INSERT IRB NAME HERE>, the sponsor of this research (NHLBI), and the Data Coordinating Center for the study may review your research and/or medical records for the purposes of verifying research data, and will see personal identifiers. However, identifying information will not appear on records retained by the sponsor, with the exception of the date of birth, subject initials, and treatment/service dates. You will not be personally identified in any reports or publications that may result from this study. There is a separate section in this consent form that you will be asked to sign which details the use and disclosure of your protected health information.

A description of this clinical trial will be available on <a href="www.clinicaltrials.gov">www.clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## PERMISSION TO RELEASE PERSONAL HEALTH INFORMATION

Authorization for Use and Disclosure of Health Information for Research Purposes

We understand that information about you and your health is personal, and we are committed to protecting the privacy of that information. Federal law requires us to get your permission to use your protected health information for this study.

Protected health information includes all information about you collected during the research study for research purposes and the information about you in medical records that is related to the research study. The information collected may include your name, date of birth, address, social security number, and results of all the tests and procedures done during the study.

If health information about you is required, the reviewers may need your entire medical record.

## USE AND DISCLOSURE COVERED BY THIS AUTHORIZATION

Who will disclose, receive, and/or use the information? The following people and organizations may disclose, use, and receive the information, but they may only use and disclose the information to the other parties on the list, to you or your legally responsible person, or as otherwise permitted or required by law.

- Investigator (study doctor), research coordinator, members of the research staff, and the Study Sponsor.
- Your study records and your entire medical record, including your personal health information may be inspected by regulatory authorities in the United States, such as the Food and Drug Administration (FDA), clinical monitor or auditor, any people or companies contracted by the sponsor (NHLBI), the Data Coordinating Center, or by <INSTITUTION> or the <INSERT IRB>. These reviews are done to check on the quality of the study.
- Members of the hospital's administrative staff who are responsible for administering clinical trials and other research activities

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

You may ask the study doctor to see and copy your personal health information related to the study. You may ask the study doctor to correct any study related information about you that is wrong. This permission to share your personal health information will expire ten years after the end of the study. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

<Insert Investigator Name, Address, Telephone number>

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you may not be able to continue to take part in the study. This is because the study staff and/or study doctor would not be able to collect the information needed to evaluate the study procedure.

The study doctor and study staff will make every effort to keep your personal health information private. But after the study staff or the study doctor share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

## IN CASE OF INJURY

If you suffer any injury as a result of taking part in this research study, please understand that nothing has been arranged to provide free treatment of the injury or any other type of payment for the injury. However, all needed facilities, emergency treatment and professional services will be available to you, just as they are to the community in general. You or your insurance provider will have to pay for those services just like any other medical care. You should report any injury to Dr. \_\_\_\_\_\_ at <INSERT principal investigator's name and phone number here> and to <INSERT IRB name and phone number here>. You will not give up any of your legal rights by signing this consent form.

### STUDY COST

All testing and services done that would not have been done but for your taking part in the study will be provided at no cost. You (or your insurance) are responsible for all other costs that are part of your usual medical care and that would have been done regardless of your enrollment in the study. If your health

insurance or Medicare requires any co-payment, co-insurance or deductible associated with your usual medical care, you will be responsible for making the payment.

You will not be paid for taking part in this study <IF SITE HAS ABILITY TO PROVIDE REIMBURSEMENT FOR PARKING FROM THE SITE BUDGET THIS CAN BE INCLUDED HERE>. If you received a bill that you believe is related to your taking part in this research study, please contact <INSERT SITE CONTACT INFO HERE> with questions.

## **QUESTIONS**

If you have questions about this clinical study or would like more specific information, you may contact the principal investigator <INSERT INVESTIGATOR NAME and 24-HOUR CONTACT NUMBER>. If you have any questions about your rights as a research study participant, you may contact the <INSERT IRB NAME AND CONTACT INFO HERE>.

### **SIGNATURES**

Sign below only if you understand the information given to you about this research study and choose to take part. Please make sure that any questions have been answered and that you understand what is being asked of you in this research study. If you have any questions or concerns about your rights as a research subject, call the <INSERT IRB NAME AND CONTACT NUMBER HERE>. If you decide to take part in this research study, a copy of this signed consent form will be given to you.

| Printed Name of Subject or Legally Authorized Representat | tive | |
|---|---|---|
| Signature of Subject or Legally Authorized Representative | Date | Time (am/pm or 24 hr) |
| I have fully explained the procedures, identifying those, wh<br>their purpose. I have asked whether or not any questions has<br>answered these questions to the best of my ability. | | |
| Printed Name of Person Obtaining Informed Consent | | |
| Signature of Person Obtaining Informed Consent | Date | Time (am/pm or 24 hr) |

#### OPTIONAL BLOOD AND TISSUE DONATION

In addition to the main part of the research study, there is an optional part of the research. You can participate in the main research without agreeing to take part in this optional research.

You have the choice of allowing us to collect additional blood samples research analysis described in the consent at a research storage laboratory facility (Biorepository Core-BRC) to be used to help further understand how stem cells function. If you agree to participate, your samples will be shipped to Dr. Doris Taylor at the BRC located at the Texas Heart Institute in Houston, Texas.

Dr. Taylor and her colleagues will use standardized processes and procedures to study which types of stem cells and related proteins might best help in the treatment of cardiovascular diseases. The remainder of the samples will be stored for future research. It is important that you know these samples: 1) will be used for research purposes only (not for profit); 2) will be stored by the BRC for up to ten years without personal identifying information, meaning it would not include any information such as your name, address, or other data that could be easily used to identify you; and 3) will be shared with researchers who will conduct studies to improve our understanding of the effects of cell therapies. Only qualified researchers will have access to the samples and data at a later date. No future studies will happen unless the investigators requesting your samples receive approval from the Institutional Review Board (IRB) that oversees their work. The purpose of the IRB is to protect the rights of participants in research studies. If for any reason you withdraw or are excluded from the study and you have consented to donate your remaining blood and tissue samples, the research team will discuss with you your options; including the possible withdrawal of consent to donate the samples. Samples will be destroyed after 10 years.

It is unlikely that these studies will have a direct benefit to you, your heirs or devisees. The results of these tests will not have an effect on your care and will not be provided to you. To avoid potential discrimination from your employer or your medical insurance, neither your doctor nor you will receive results of these future studies, nor will the results be put in your health record.

Although we have systems in place to protect your identity, there is always a potential risk of loss of confidentiality. Sometimes blood and tissue samples are used for genetic research about diseases that are passed on in families. Even if your samples are used for this kind of research, the results will not be put in your health records and every effort will be made to keep your identity confidential. The study investigator <INSERT INVESTIGATOR NAME HERE> does not have ownership or proprietary interest in these samples. There are no plans to provide financial compensation to you, your heirs or devisees (those listed in your will).

If you do not wish to donate any blood or tissue samples to the BRC, it will not affect your eligibility for taking part in this study.

Please review the sample requests below and indicate your preferences regarding the optional collection and storage of your blood and tissue samples for future research studies.

# **COLLECTION OF BLOOD SAMPLES**

| <ul> <li>Blood samples – (each draw is about 1.5 tablespoons) will be collected at:</li> <li>Study product injection visit- before study product delivery</li> </ul> |
|---|
| <ul> <li>Study product injection visit- before study product delivery</li> <li>Day after product injection –prior to discharge from hospital</li> </ul> |
| <ul> <li>During three follow up visits (week 1, month 1, and month 6) - these samples will be collected during the blood draws already scheduled for the main study.</li> </ul> |
| ☐ I do voluntarily consent to donate additional blood samples to the biorepository. |
| ☐ I do not consent to donate additional blood samples to the biorepository. |
| COLLECTION OF TISSUE SAMPLES |
| <b>Explanted Heart-</b> In the event of death or a heart transplant, the researcher requests your permission to do an examination of your old heart so that researchers can gain a better understanding of the consequences of cell transfer. |
| <ul> <li>I do voluntarily consent to donate my old heart in the event of my death or following my heart transplant to the biorepository.</li> <li>I do not consent to donate my old heart upon my death or transplant to the biorepository.</li> </ul> |
| USE AND STORAGE OF SAMPLES FOR FUTURE RESEARCH |
| Future research studies (e.g. study of proteins) about cardiovascular diseases. |
| Yes, I <u>agree</u> for my samples to be used and stored for <i>cardiovascular research</i> . |
| No, I do not agree for my samples to be used and stored for <i>cardiovascular research</i> . |
| ☐ Did not consent to any sample collection (in previous section) |
| Genetic research studies (e.g. using DNA and RNA) about cardiovascular diseases. |
| Yes, I <u>agree</u> for my samples to be used and stored for <i>genetic</i> studies of cardiovascular disease. |
| No, I do not agree for my samples to be used and stored for genetic studies of cardiovascular disease. |
| ☐ Did not consent to any sample collection (in previous section) |
| De-identified information about me (e.g. age, smoking history, etc.) may be included in a data set that is available to qualified researchers outside the study. |
| Yes, I <u>agree</u> for de-identified information about me to be included in a data set. |
| No, I do not agree for de-identified information about me to be included in a data set. |
| Did not consent to any sample collection (in previous section) |

| preferences for the collection of your specimens as well as the | | 1 |
|---|---|---|
| Printed Name of Subject or Legally Authorized Representative | | |
| Signature of Subject or Legally Authorized Representative | Date | Time (am/pm or 24 hr) |
| I have fully explained the procedures, identifying those, which purpose. I have asked whether or not any questions have arisen questions to the best of my ability. | | |
| Printed Name of Person Obtaining Informed Consent | | |
| Signature of Person Obtaining Informed Consent | Date | Time (am/pm or 24 hr) |
| This study <insert approval="" here="" irb="" number=""> has IRB HERE&gt; of <insert here="" institution="" name="">. Fo or to report a research-related injury, call the IRB at <insert< td=""><td>r any questi</td><td>ions about research subject's rights,</td></insert<></insert></insert> | r any questi | ions about research subject's rights, |